CLINICAL TRIAL: NCT03370237
Title: Reliability of a Diabetic Foot Ulcer Risk Stratification and Referral Algorithm
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: St. Joseph's Healthcare Foundation (Other)
Responsible Party: Principal Investigator, Elisabeth Harvey, Adjunct Associate Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 30
Record Dates: First submitted 2017-12-07; First posted 2017-12-12 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Foot Ulcer, Diabetic
Keywords: Diabetic foot ulcer; type 2 diabetes; foot ulcer risk
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this research study is to validate the St Joseph's Health Care Harmonized Foot Ulcer Assessment and Stratification tool using inter-rater reliability technique to determine if the score would consistently be reproducible by examiners of different role (Nurse Practitioner, Family physician, Registered Nurse and Resident). A validated assessment tool allows collecting better quality data with high comparability which enhances quality of foot care and increases the credibility of the tool.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a chronic disease characterized by the human body's inability to maintain appropriate blood glucose levels ( Buse et al. 2011). When inadequately managed, diabetes results in poor glycemic control, which, if prolonged, results in diabetes-related complications (Stratton et al. 2000). Diabetes is the major cause of blindness, kidney failure, and non-traumatic amputation in Canadian adults (PHAC, 2011). Foot ulcers are the major causes of amputations. Foot ulcers arise from poor circulation associated with peripheral vascular disease and neuropathy, injury and infections. Diabetes affects circulation and immunity, and over time the sensory nerves in the hands and feet may be damaged.

There are more than 2.4 million Canadians living with diabetes, of which 1.2 million of them live in Ontario (MHLTC). Diabetes is the leading cause of non-traumatic lower limb amputation in Canadian adults, associated with approximately 70% of amputations performed in hospital. Compared to the general population, Canadian adults with diabetes are over 20 times more likely to undergo non-traumatic lower limb amputations, 85% of which are preceded by a foot ulcer (PHAC, 2011 and Singh et al.,2005). According to a recent report (CDA, 2016) commissioned by the Canadian Diabetes Association (CDA), of the 1.53 million people with diabetes in Ontario, between 16,600 and 27,600 were expected to have a diabetes foot ulcer in 2015. Of these, nearly 2,000 were expected to need to have a lower limb amputated as a result of their condition and those amputations are associated with almost 800 premature deaths. In Ontario, diabetic foot ulcers (DFU) currently impose direct health-care costs of between $320-400 million and indirect costs of between $35-60 million (Hopkins et al.,2015).

Strong evidence shows that up to 85% of diabetic foot amputations can be prevented, supporting the benefits of early recognition of diabetes-related foot complications (CDA, 2013). Furthermore, timely assessment, referral, and provision of evidence-informed foot care are cost saving for the healthcare system. Use of a standardized diabetic foot assessment tool is required to ensure consistent approach to risk recognition and provide a framework for care. In response to the need for a tool that facilitates a consistent and standard screening procedure, the Primary Care Diabetes Support Program (PCDSP) at St. Joseph's Health Care, London, Ontario developed an evidence based, multi-disciplinary foot ulcer assessment tool. The SJHC harmonized foot ulcer assessment tool was developed to aid in the early detection of diabetic foot problems and to ensure prompt referral to the right foot care provider for appropriate treatment, thereby improving outcomes of the diabetic foot.

ELIGIBILITY:
Inclusion Criteria:

Patients with type 2 diabetes older than 18, living with diabetes for more than ten years and consented were included in the study as patient participants.

Care providers including family doctors, nurse practitioners, nurses and residents who provider diabetes care was including as care provider participants

Exclusion Criteria:

Patients with previous transfemoral or transtibial amputation or diagnosed with dementia or inability to speak English were excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with type 2 diabetes who have received diabetes care at the primary care diabetes support program in London Ontario, Canada.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-09-22 (Actual); Study Completion 2017-09-22 (Actual)

PRIMARY OUTCOMES:
Diabetic foot ulcer risk score | on examination day
  The Diabetic Foot Ulcer Assessment tool used in this study has five scores (categories) ranging from 0(low risk) to 3A (high risk). The higher the score is the higher the risk for diabetic foot ulcer. Each care provider assessed participating patients for foot ulcer and assigned a score for each. The five scores are 0, 1,2A,2B and 3A.

SECONDARY OUTCOMES:
Raters' level of confidence | On examination day
  Raters (care providers) level of confidence in using the tool to assess diabetic foot and plan appropriate follow up

CONTACTS AND LOCATIONS:
Overall Officials: Betty Harvey, Principal Investigator — Western University and St Joseph's Health Care London
Locations (1):
- SJHC Primary Care Diabetes Support Program SJHC Family Medical and Dental Centre, London, Ontario, Canada

REFERENCES:
- [Background] Buse JB, Polonsky KS, Burant CF. Type 2 diabetes mellitus. In: Kronenberg HM, Melmed S, Polonsky KS, Larsen PR. Williams Textbook of Endocrinology. 12th ed. Philadelphia, PA: Saunders Elsevier; 2011
- [Background] Stratton IM, Adler AI, Neil HA, Matthews DR, Manley SE, Cull CA, Hadden D, Turner RC, Holman RR. Association of glycaemia with macrovascular and microvascular complications of type 2 diabetes (UKPDS 35): prospective observational study. BMJ. 2000 Aug 12;321(7258):405-12. doi: 10.1136/bmj.321.7258.405. PMID 10938048
- [Background] Public Health Agency of Canada. Diabetes in Canada: Facts and Figures from a Public Health Perspective. Ottawa; 2011.
- [Background] Ministry of Health and Long Term Care. Diabetes Management Strategy. Chapter 3 Section 3.03
- [Background] Singh N, Armstrong DG, Lipsky BA. Preventing foot ulcers in patients with diabetes. JAMA. 2005 Jan 12;293(2):217-28. doi: 10.1001/jama.293.2.217. PMID 15644549
- [Background] Canadian Diabetes Association : Impact of offloading devices on the cost of diabetic foot ulcers in Ontario, http://www.diabetes.ca/publications-newsletters/advocacy-reports/impact-of-offloading-devices Accessed on Sep 11 2016
- [Background] Hopkins RB, Burke N, Harlock J, Jegathisawaran J, Goeree R. Economic burden of illness associated with diabetic foot ulcers in Canada. BMC Health Serv Res. 2015 Jan 22;15:13. doi: 10.1186/s12913-015-0687-5. PMID 25608648
- [Background] Canadian Diabetes Association Clinical Practice Guidelines Expert Committee; Booth G, Cheng AY. Canadian Diabetes Association 2013 clinical practice guidelines for the prevention and management of diabetes in Canada. Methods. Can J Diabetes. 2013 Apr;37 Suppl 1:S4-7. doi: 10.1016/j.jcjd.2013.01.010. Epub 2013 Mar 26. No abstract available. PMID 24070961